CLINICAL TRIAL: NCT01401114
Title: Drug Use Investigation of Wellnara Tablet
Brief Title: Wellnara Post-marketing Surveillance in Japan
Acronym: WELLNARA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15041
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Wellnara; Postmenopausal osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Drug (incl. Placebo)
  Interventions: Drug: E2/LNG oral (Wellnara, BAY86-5029)

INTERVENTIONS:
Drug: E2/LNG oral (Wellnara, BAY86-5029) — Patients in daily life treatment receiving Wellnara for postmenopausal osteoporosis

SUMMARY:
This study is a regulatory post marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Wellnara for postmenopausal osteoporosis. The objective of this study is to assess safety and efficacy of using Wellnara in clinical practice. A total 400 patients will be recruited and followed 3 years since starting Wellnara administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Wellnara for postmenopausal osteoporosis

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who have received a prescription of Wellnara on the basis of the decision of the treating gynecologist. The study is expected to collect data of 400 patients in about 80 gynecological practices in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2009-03; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in subject who received Wellnara | After Wellnara administration, up to 3 years

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation with baseline data (such as demographic data, concomitant disease) and dose of Wellnara | At baseline and after Wellnara administration, up to 3 years
Effectiveness evaluation assessment by the three rank scales: improvement, not changed, and worse | At baseline and after Wellnara treatment, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan